CLINICAL TRIAL: NCT02161003
Title: Therapeutic Effect of Stem Cells in Fecal Incontinence in Children After Posterior Sagittal Ano-rectoplasty
Brief Title: Stem Cells Therapy for Fecal Incontinence in Children After Posterior Sagittal Ano-rectoplasty
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Collaborators: Cairo University (Other); Ain Shams University (Other); Affiliated Hospital to Academy of Military Medical Sciences (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Sayed Bakry, Associate Professor - Consultant of Isolation and Culturing of Stem Cells, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Azhar52980070; Azhar52980070 (Other Grant/Funding Number: Al Azhar University)
Record Dates: First submitted 2014-05-09; First posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Fecal Incontinence
Keywords: Fecal Incontinence; Posterior Sagittal Ano-rectoplasty; Mesenchymal Stem Cell
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stem Cells Isolation (Experimental): Stem cell isolation technique and Stem Cells Injection Technique The method of isolation of MSC from bone marrow will be carried out using the Ficoll-Paque technique for the isolation of mononucleated cells followed by the separation of MSC by adherence to plastic. Finally, the cells will be resuspended and counted using a hemocytometer.
  Mononucleated cells will be cultured and incubated at 37°C in an atmosphere of 95% relative humidity and 5% CO2.
  Interventions: Procedure: Stem Cells Injection Technique; Procedure: Stem Cell Isolation

INTERVENTIONS:
Procedure: Stem Cells Injection Technique — Injection of MSCs for the treatment of anal sphincter insufficiency is a potential alternative therapy for imperforate anus patients who have undergone primary PSARP with post-operative FI. In this study a single dose of 1.2 ml MSC will be divided into 12 part of 0.1ml of MSC, doses will be injected into the anal sphincter all around in 12 injection sites according to the clock meridian under general anesthesia without giving muscle relaxant.
Procedure: Stem Cell Isolation — From the upper posterior iliac crest 10 ml bone marrow sample will be extracted from patients using a heparinized syringe, under general anesthesia, in a suitable clean operation room.

SUMMARY:
The problem of the incontinence imposes considerable strain on the child and their parents. These patients suffer from a long-life handicap and they need support and follow-up. The cost associated with these diseases has clearly been illustrated to be a major component in the healthcare spending picture, may be adding hundreds of thousands of dollars to healthcare cost, as well as loss of productivity in the work force. Fecal incontinence treatment has been a difficult challenge for surgeons for several generations until now the current traditional surgical result is unsatisfactory. Mesenchymal Stem Cells injection may represent a new attractive treatment option for anal sphincter lesions. Moreover, experimental injury of muscle of anal sphincter in rats has been successfully treated with stem cells injections. In this study, the investigators will shed more light on the ability of Mesenchymal Stem Cells to induce myogenesis and regenerate anal Sphincter of patients with fecal incontinence. It will be very useful to many Egyptian patients.

DETAILED DESCRIPTION:
A stem cell is capable of forming various tissue under definite signals received from the body. Stem cell research in animals has been an ongoing program in the west with fruitful results. Current challenges with the use of stem cells in clinical practice will be solve the many unanswered queries. To study the potential therapeutic effects of local Mesenchymal Stem cell injection in children presenting with fecal incontinence (FI) after posterior sagittal ano-rectoplasty (PSARP) operation for high imperforate anus. Children whom suffering from FI after PSARP for high imperforate anus will included in this study. Autologous MSC from the upper posterior iliac crest bone marrow sample will be extracted from patients under general anesthesia, in a suitable clean operation room. Will be Cultured and injected into the external anal sphincter defect using direct pena stimulator or ultra sound guidance. Then followed up for 180 days post injection, to assess the ability of mesenchymal stem cells to induce myogenesis of the anal Sphincter of patients with FI after PSARP.

ELIGIBILITY:
Inclusion Criteria:

Male Childern Ages: above 2 Years old.

Patient with FI. After PSARP repair of high imperforate anus.

Absence of parasitic and infective bacterial growth after Stool analysis and stool culture.

-

Exclusion Criteria:

Any degree of Spinal cord injury, systemic, neuronal paralysis or sacral agenesis.

Absence of muscle activity detected by EMG.

Ano-rectal disorders such as tumors, fissures, anal or rectal prolapse, and rectocele.

Positive stool culture resistant to preoperative oral antibiotic therapy.

Previous injection of bulking agents at the level of sphincter.

Immunocompromise patient.

Previous adverse reaction to anesthesia.

Ages: 2 Years to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Main outcome measures | 24 Weeks
  Incontinence Score

SECONDARY OUTCOMES:
Assessment of Clinical Parameters | 24 Weeks
  This Including:
  Clinical Assessment. Continence score.
Clinical Assessment | 12 Weeks
  Maximum dry interval per day will be measured after injection at day 1, 30 and 90.
Clinical Assessment | 24 Weeks
  MRI pelvic floor muscles study will be done after 90 days post injection.
Assessment of Urinary sphin Assessment of Urinary Sphincter (Electrophysiology Study) | 48 Weeks
  EMG study will be done after 90, 180 days post injection.

CONTACTS AND LOCATIONS:
Overall Officials: Abdel-Wahab El-Okby, MD, Principal Investigator — Al-Azhar University; Naglaa Ali Gadallah, MD, Study Chair — Ain Shams University; Sayed Bakry, PhD, Study Director — Al-Azhar University; Refaat El-Badawy, MD, Study Chair — Al-Azhar University; Hala Gabr, MD, Study Chair — Cairo University; Wael Wael Abu El Khier, MD, Study Chair — Military Academy; Anthony Atala, MD, Study Chair — Director of the Wake Forest Institute for Regenerative Medicine; Mostafa Elbahrawy, MSc, Study Chair — Al-Azhar University
Locations (1):
- Pediatric Surgery Outpatients Clinics - Al Hussien Hospital, Madīnat an Naşr, Cairo Governorate, Egypt